CLINICAL TRIAL: NCT06532253
Title: Long-term Safety Bucket Trial with NVDX3, an Osteogenic Implant of Human Allogenic Origin.
Brief Title: Long-term Safety Trial with NVDX3
Acronym: X3LTFU
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novadip Biosciences (Industry)
Collaborators: PrimeVigilance (Industry); Data Investigation Company Europe (DICE) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVDX3-CLN0X
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-07

CONDITIONS: Distal Radius Fractures; Degenerative Lumbar Spondylolisthesis
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NVDX3 implant (Experimental): NVDX3 implant is a sterilized, dry powder. The total administered quantity of NVDX3 implant depends on the bone defect size/intervertebral disc space.
  Interventions: Drug: NVDX3

INTERVENTIONS:
Drug: NVDX3 — NVDX3 is implanted during a single surgical intervention, that took place in the core trials (refer to NCT05961956 and NCT05987033)

SUMMARY:
An study evaluating the long-term safety of all patients previously treated with NVDX3.

DETAILED DESCRIPTION:
An study evaluating the long-term safety of all patients previously treated with NVDX3 (referred to as the "core NVDX3 trial"). All patients having signed the ICF enter the long term follow-up study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient being implanted with NVDX3.
2. Previously participated to one of the NVDX3 core clinical trials.
3. Patient accepts to comply to a yearly follow-up safety visit for 10 additional years
4. Patient has understood and accepted to participate in the long-term follow-up study by signing the informed consent.

Exclusion Criteria:

No exclusion criteria are applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2036-03 (Estimated); Study Completion 2036-03 (Estimated)

PRIMARY OUTCOMES:
Long-term safety of the NVDX3 implant | Between screening (V0) and 120 months post-core study (V10)
  Description of all SAEs, NVDX3 related AEs and AE of special interest

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Gerich, MD, Principal Investigator — Centre Hospitalier du Luxembourg
Locations (1):
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg